CLINICAL TRIAL: NCT00533260
Title: A Non-interventional Naturalistic Project to Investigate the Effect of the Use of SMS Text Service on Treatment Adherence in Patients Treated With Seroquel®
Brief Title: A Non-interventional Naturalistic Project to Investigate the Effect of the Use of SMS Text Service on Treatment Adherence in Patients Treated With Seroquel® (Quetiapine)
Acronym: SEQUEL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-NNL-SER-2007/1
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: Patients with a manic episode or patients diagnosed with schizophrenia , patients who are being treated with quetiapine and are on a stable dosing regime
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The basic hypothesis of this trial is that forgetfulness and failure to establish a routine that facilitates medication adherence are prominent reasons for non-adherence. Daily use of the SMS text messages is designed to enhance patient adherence with medication by promoting daily routine and demonstrate the feasibility of using SMS technology within normal clinical practice in The Netherlands.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* The subjects should be considered eligible for this trail according to the physician:

  1. Patients with a diagnose of schizophrenia or bipolar disorder with a recent manic episode
  2. Patients who are being treated with quetiapine and are on an effective dose according to the Core Data Sheet; for schizophrenia between 300 and 450 mg (maximum 750 mg) and bipolar disorder between 400 and 800 mg.
  3. Patients who consent to make the coded data available to AstraZeneca; provision of written informed consent
  4. Considered eligible for this study and able to understand and comply with the requirements of the study according to the physician
  5. In possession of a private mobile phone and capable of using this mobile phone to send SMS text messages

Exclusion Criteria:

* Subjects who, in the opinion of the Physician, pose an imminent risk of suicide or a danger to themselves or others are excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were considered for participation were patients who were being treated with quetiapine according to the Core Data Sheet and who were on a stable dosing regime. They could have been patients with schizophrenia or patients experiencing a manic episode associated with a bipolar disorder. Quetiapine was administered to the patients in regular practice.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: N van Schayk, Study Director — AstraZeneca
Locations (35):
- Netherlands (35):
  - Research Site, Almelo
  - Research Site, Alphen Aan de Rigjn
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Arnhem
  - Research Site, Bennebroek
  - Research Site, Beverwijk
  - Research Site, Bosch en Duin
  - Research Site, Brummen
  - Research Site, Brunssum
  - Research Site, Doetichem
  - Research Site, Druten
  - Research Site, Ede
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Heerde
  - Research Site, Helmond
  - Research Site, Hoofddorp
  - Research Site, IJmuiden
  - Research Site, Leeuwarden
  - Research Site, Maastricht
  - Research Site, Nijbroek
  - Research Site, Nijmegen
  - Research Site, Oegstgeest
  - Research Site, Raalte
  - Research Site, Roermond
  - Research Site, Schagen
  - Research Site, Steenwijk
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Venray
  - Research Site, Vlaardingen
  - Research Site, Voorhout
  - Research Site, Weert
  - Research Site, Wolfheze